CLINICAL TRIAL: NCT03036904
Title: Phase I Study of Venetoclax Plus DA-EPOCH-R for the Treatment of Aggressive B-Cell Lymphomas
Brief Title: Study of Venetoclax Plus DA-EPOCH-R for the Treatment of Aggressive B-Cell Lymphomas
Acronym: V+DA-EPOCH-R
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry); Massachusetts General Hospital (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1607017413
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Diffuse Large B-Cell Lymphoma; High Grade B-Cell Lymphoma
Keywords: venetoclax; dose-adjusted EPOCH-R; aggressive B-Cell lymphoma; Lymphoma; Non-Hodgkin lymphoma; Diffuse large B-cell lymphoma; Double hit lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma; Lymphoma, Non-Hodgkin | interventions — venetoclax; Rituximab; Etoposide; etoposide phosphate; Vincristine; Cyclophosphamide; Prednisone; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax plus DA-EPOCH-R (Experimental): Venetoclax will be given in conjunction with 6 cycles of DA-EPOCH-R (doxorubicin hydrochloride, etoposide, vincristine sulfate, cyclophosphamide, prednisone, rituximab). The dosing schedule and regimen for DA-EPOCH-R will follow established protocols. Venetoclax will be administered days 1-10 of each 21-day cycle, with the exception of cycle 1, during which venetoclax dose will commence on day 3 and continue through day 12, so as to clarify attribution of any observed TLS and/or infusion reactions, and minimize tumor lysis syndrome (TLS) risk.
  Interventions: Drug: Venetoclax; Drug: Rituximab; Drug: Etoposide; Drug: Vincristine Sulfate; Drug: Cyclophosphamide; Drug: Prednisone; Drug: Doxorubicin Hydrochloride

INTERVENTIONS:
Drug: Venetoclax — Venetoclax will be administered orally on days 3-12 in cycle 1, and days 1-10 with all subsequent cycles except dose level -1. If dose level -1 is required, venetoclax will be administered on days 3-7 in cycle 1 and 1-5 with subsequent cycles.
  Other Names: Venclexta
Drug: Rituximab — Rituximab will be administered as an IV infusion at 375 mg/m2 on day 1 of each cycle of DA-EPOCH-R, immediately prior to the start of chemotherapy. Oral pre-medication 650 mg of acetaminophen and 50-100 mg diphenhydramine hydrochloride will be administered 30 to 60 minutes prior to starting each infusion of rituximab. The first rituximab infusion should be started at 50 mg/hr, and increased in 50-mg/hr increments every 30 minutes to a maximum rate of 400 mg/hr. If this rate of escalation is well tolerated the second and subsequent infusions can begin at a rate of 100 mg/hr and increase in 100 mg/hr increments every 30 minutes to a maximum of 400 mg/hr. CAUTION: DO NOT ADMINISTER AS AN INTRAVENOUS PUSH OR BOLUS.
  Other Names: Rituxan; IDEC-C2B8; chimeric anti-CD20 monoclonal antibody
Drug: Etoposide — Etoposide will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: VP-16; VePesid; etopophos; toposar
Drug: Vincristine Sulfate — Vincristine Sulfate will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: LCR; VCR
Drug: Cyclophosphamide — Cyclophosphamide will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: cytoxan
Drug: Prednisone — Prednisone will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. Prednisone will be given orally.
  Other Names: Deltasone; Orasone; Paracort; Cortan
Drug: Doxorubicin Hydrochloride — Doxorubicin Hydrochloride will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: Hydroxydaunomycin Hydrochloride; Hydroxydoxorubicin Hydrochloride

SUMMARY:
This is a phase I, open label, single-arm, multi-center, dose-finding study of venetoclax in combination with DA-EPOCH-R in patients with aggressive B-Cell Lymphomas.

DETAILED DESCRIPTION:
This clinical trial is for men and women with aggressive B-Cell Lymphomas which includes:

* Diffuse large B-cell lymphoma (DLBCL),
* B-cell lymphoma unclassifiable with intermediate features between DLBCL and Burkitt Lymphoma (BL),
* High grade B-cell lymphoma (HGBCL),
* Transformed indolent NHL (TiNHL). The aggressive B-cell lymphomas enrolling on this study have been recognized to have a poor prognosis with the use of conventional chemoimmunotherapy. DA-EPOCH-R is an alternative highly effective chemoimmunotherapy platform for these lymphomas and may serve as an optimal chemotherapy backbone for the incorporation of novel agents such as venetoclax.

The Bcl-2 protein plays a significant role in the regulation of cell death in malignant cells. Overexpression of Bcl-2 family proteins is associated with chemo-resistance of a broad variety of cancers, and BCL2 abnormalities are common in aggressive B-cell Lymphomas. Venetoclax is a highly selective Bcl-2 family protein inhibitor that binds to Bcl-2 family proteins to potentially overcome resistance and enhance responses to therapy. This study has been designed to evaluate the safety and preliminary efficacy of venetoclax in combination with DA-EPOCH-R.

Subjects will receive venetoclax in conjunction with six 21-day cycles of DA-EPOCH-R. Dosing for DA-EPOCH-R will follow established protocols. Venetoclax will be administered on days 3 through 12 during cycle 1 and days 1 through 10 of each subsequent cycle. Following completion of therapy, subjects will be followed every three months for up to two years. Subjects removed from study due to toxicity will be followed until resolution or stabilization of the toxicity.

ELIGIBILITY:
Inclusion criteria:

* Adults age 18-80 years
* Histologically confirmed, biopsy-proven diagnosis of DLBCL, BCLu, HGBCL, or TiNHL.

Richter's transformation from Chronic Lymphocytic Leukemia (CLL) is not eligible.

* Subjects with DLBCL, BCLu, HGBCL NOS, or HGBCL with translocations of MYC and BCL2 and/or BCL6, must have had no prior chemotherapy for lymphoma. Steroids for palliation prior to enrollment are allowed.
* Subjects with TiNHL are eligible if they have received no prior cytotoxic chemotherapy for lymphoma. Steroids, rituximab, and external beam radiation therapy as prior therapy for indolent lymphoma is allowed.
* Ann Arbor stage II-IV disease (Stage I primary mediastinal B-cell lymphoma will also be eligible)
* Ability to provide signed Informed Consent Form
* Ability and willingness to comply with the requirements of the study protocol
* Measureable disease (defined as at least 1.5 cm in diameter).
* Adequate organ and bone marrow function:
* Absolute neutrophil count (ANC) at least 1,000/mm3
* Platelet count at least 100,000/mm3.
* Total bilirubin at most1.5 x the upper limit of the normal range (ULN), except Gilbert's disease
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) at most 3 x ULN.
* Calculated creatinine clearance at least 30 mL/min.

Exclusion criteria:

* Known hypersensitivity to any of the study drugs
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will also be excluded, unless the malignancy has been in remission without treatment for at least 2 years prior to enrollment.
* Known CNS involvement at diagnosis
* Richter's transformation from CLL
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal)
* Major surgery within 3 weeks prior to the start of study treatment
* Infection with human immunodeficiency virus (HIV)
* Women who are pregnant or lactating
* Female patients who are not surgically sterile or postmenopausal (for at least 1 year) must practice at least one of the following methods of birth control throughout the duration of study participation and for at least 3 months after study treatment:
* Total abstinence from sexual intercourse
* A vasectomized partner
* Hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) that started at least 3 months prior to study drug administration
* Double-barrier method (condom plus diaphragm or cervical cup with spermicidal contraceptive sponge, jellies, or cream)
* Non-vasectomized male patients must comply with at least one of the following methods of birth control throughout the duration of study participation and for at least 3 months after study treatment:
* A partner who is surgically sterile or postmenopausal (for at least 1 year) or who is taking hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) for at least 3 months prior to study drug administration
* Total abstinence from sexual intercourse
* Double-barrier method (condom plus diaphragm or cervical cup with spermicidal, contraceptive sponge, jellies, or cream)
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase
* Subjects with positive HBV core antibody or surface antigen are eligible as long as they have an undetectable HBV DNA PCR, and receive concurrent antiviral therapy with entecavir, tenofovir, or lamivudine, and continued for a minimum of 6 months after completion of therapy.
* Active hepatitis C (defined as a positive HCV viral load)
* Chronic use of moderate or strong CYP3A4 modulators (inhibitor or inducer) or any other prohibited medications. A washout period of 7 days is required prior to venetoclax dosing if a prohibited medication is discontinued.
* Chronic use of a P-gp inhibitor, or a P-gp substrate with a narrow therapeutic index. A washout period of 7 days is required prior to venetoclax dosing if a prohibited medication is discontinued.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Determination of the maximal tolerated dose (MTD) | Approximately 24 months
  Determination of the maximal tolerated dose (MTD)
Determination of dose limiting toxicity (DLT) | Approximately 24 months
  Determination of dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Define incidence and severity of adverse events, defined according to CTCAE v 4.0. | Approximately 24 months
  Define incidence and severity of adverse events, defined according to CTCAE v 4.0.
Overall response rate | Approximately 24 months
  Overall response rate
Complete response rate | Approximately 24 months
  Complete response rate
Event-free survival | Approximately 24 months
  Event-free survival
Progression Free Survival | Approximately 24 months
  Progression Free Survival
Overall survival | Approximately 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: John P. Leonard, M.D., Study Chair — Weill Medical College of Cornell University; Jeremy S. Abramson, M.D., Study Chair — Massachusetts General Hospital; Sarah Rutherford, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (6):
- United States (6):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Weill Cornell Medicine, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutherford SC, Abramson JS, Bartlett NL, Barta SK, Khan N, Joyce R, Maddocks K, Ali-Shaw T, Senese S, Yuan Y, Westin J, Leonard JP. Venetoclax with dose-adjusted EPOCH-R as initial therapy for patients with aggressive B-cell lymphoma: a single-arm, multicentre, phase 1 study. Lancet Haematol. 2021 Nov;8(11):e818-e827. doi: 10.1016/S2352-3026(21)00273-8. Epub 2021 Oct 8. PMID 34634256